CLINICAL TRIAL: NCT05385770
Title: A Multicentre, Randomized, Double-blind Study to Evaluate and Compare the Efficacy and Safety of 8-week Treatment With AZM and AML Combined and Alone in Mild-to-moderate Essential Hypertensive Subjects
Brief Title: Study to Evaluate and Compare the Efficacy and Safety of AZM and AML Combined and Alone in Mild-to-moderate Essential Hypertensive Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-L05-301
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Single-blind Run-in period, Double-blind Treatment period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- AZM Xmg (Active Comparator): 1. AZM Xmg (4 weeks) Non-responder -> AZM Xmg (8 weeks)
  Interventions: Drug: AZM X mg
- AZM X'mg (Active Comparator): 1. AZM X'mg (4 weeks) Non-responder -> AZM X'mg (8 weeks)
  Interventions: Drug: AZM X' mg
- AML Ymg (Active Comparator): 1. AML Ymg (4 weeks) Non-responder -> AML Ymg (8 weeks)
  Interventions: Drug: AML Y mg
- AML Y'mg (Active Comparator): 1. AML Y'mg (4 weeks) Non-responder -> AML Y'mg (8 weeks)
  Interventions: Drug: AML Y' mg
- AZM/AML X/Ymg (Active Comparator): 1. AZM Xmg (4 weeks) Non-responder -> AZM Xmg + AML Ymg (8 weeks)
  2. AML Ymg (4 weeks) Non-responder -> AZM Xmg + AML Ymg (8 weeks)
  Interventions: Drug: AZM X mg + AML Y mg; Drug: AZM X mg; Drug: AML Y mg
- AZM/AML X'/Ymg (Active Comparator): 1. AZM X'mg (4 weeks) Non-responder -> AZM X'mg + AML Ymg (8 weeks)
  2. AML Ymg (4 weeks) Non-responder -> AZM X'mg + AML Ymg (8 weeks)
  Interventions: Drug: AZM X' mg + AML Y mg; Drug: AZM X' mg; Drug: AML Y mg
- AZM/AML X/Y'mg (Active Comparator): 1. AZM Xmg (4 weeks) Non-responder -> AZM Xmg + AML Y'mg (8 weeks)
  2. AML Y'mg (4 weeks) Non-responder -> AZM Xmg + AML Y'mg (8 weeks)
  Interventions: Drug: AZM X mg + AML Y' mg; Drug: AZM X mg; Drug: AML Y' mg
- AZM/AML X'/Y'mg (Active Comparator): 1. AZM X'mg (4 weeks) Non-responder -> AZM X'mg + AML Y'mg (8 weeks)
  2. AML Y'mg (4 weeks) Non-responder -> AZM X'mg + AML Y'mg (8 weeks)
  Interventions: Drug: AZM X' mg + AML Y' mg; Drug: AZM X' mg; Drug: AML Y' mg

INTERVENTIONS:
Drug: AZM X mg + AML Y mg — tablet, single dose, QD, oral administration
  Arms: AZM/AML X/Ymg
Drug: AZM X mg + AML Y' mg — tablet, single dose, QD, oral administration
  Arms: AZM/AML X/Y'mg
Drug: AZM X' mg + AML Y mg — tablet, single dose, QD, oral administration
  Arms: AZM/AML X'/Ymg
Drug: AZM X' mg + AML Y' mg — tablet, single dose, QD, oral administration
  Arms: AZM/AML X'/Y'mg
Drug: AZM X mg — tablet, single dose, QD, oral administration
  Arms: AZM Xmg; AZM/AML X/Y'mg; AZM/AML X/Ymg
Drug: AZM X' mg — tablet, single dose, QD, oral administration
  Arms: AZM X'mg; AZM/AML X'/Y'mg; AZM/AML X'/Ymg
Drug: AML Y mg — tablet, single dose, QD, oral administration
  Arms: AML Ymg; AZM/AML X'/Ymg; AZM/AML X/Ymg
Drug: AML Y' mg — tablet, single dose, QD, oral administration
  Arms: AML Y'mg; AZM/AML X'/Y'mg; AZM/AML X/Y'mg

SUMMARY:
This is an 8-week, randomized, double-blind Phase 3, multicentre study to determine the optimal dose of AZM and AML in combination therapy and to compare efficacy and tolerability of the combined therapy to each of the monotherapy in essential hypertensive subjects who are not adequately controlled on AZM and AML monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily agree to participate in the trial and signed the written ICF, after listening to the purpose, method, and effect of clinical trial
* Male or female adult subjects (Legal minimum age of adult requirement is country specific, and requirement of current country specific regulations will be applied) below the age of 75 years, inclusive
* Subjects with mild-to-moderate essential hypertension
* Subjects who are capable of understanding and complying with protocol requirements

Exclusion Criteria:

* Subjects who have msitSBP >180 mmHg or msitDBP >110 mmHg; Subjects who have difference in the blood pressure between 3 measurements (confirmed by a second set of three measurements; 3 sitting systolic BP (sitSBP) measurements differing by more than 20 mmHg or 3 sitting diastolic BP (sitDBP) measurements differing by more than 10 mmHg)
* Secondary hypertension, Symptomatic orthostatic hypotension
* Clinically significant Electrocardiogram (ECG) abnormalities, Severe heart disease, Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically significant arrhythmia, Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
* Severe cerebrovascular disease, Known moderate or malignant retinopathy within the past 6 months; History of unexplained syncope within the prior 2 years, or a known syncopal disorder
* Significant thyroid disease, Type 1 or 2 diabetes mellitus with poor glucose control, Wasting disease, Autoimmune diseases, Connective tissue disease
* Subjects who have clinically significant laboratory abnormalities : creatinine clearance < 30 mL/min, serum creatinine > 2 mg/dL or > 200 μmol/L, serum potassium <3.5 mmol/L or > 5.5mmol/L, alanine aminotransferase or aspartate aminotransferase > 3 × upper limit normal (ULN)
* Any surgical or medical condition of the gastrointestinal tract that might significantly alter the absorption, distribution, metabolism, or excretion of the drug
* Positive for HIV, HCV Ab, and/or HBsAg
* History of drug or alcohol abuse within the past 1 year
* Subjects who are pregnant or lactating women, women suspected of being pregnant, women who wish to be pregnant during the study, or women of child-bearing potential who are not using medically acceptable methods of contraception
* Any chronic inflammatory condition needing chronic anti-inflammatory therapy, A known hypersensitivity to any main excipients and components of the investigational drugs or other drugs in the same class, Subjects who have previously experienced symptoms characteristic of angioedema during treatment with angiotensin-converting enzyme inhibitors or angiotensin II subtype 1 receptor blocker
* Subjects who have received any investigational product within 28 days prior to screening or is currently participating in another investigational study
* Subjects who are required to take excluded medications at any point during the study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 890 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
msitSBP | after 8 weeks of treatment
  msitSBP change from baseline

SECONDARY OUTCOMES:
msitDBP | after 8 weeks of treatment
  msitDBP change from baseline
msitSBP | after 4 weeks of treatment
  msitSBP change from baseline
msitDBP | after 4 weeks of treatment
  msitDBP change from baseline
Proportion of subjects achieving msitSBP < 140 mmHg and/or ΔmsitSBP ≥ 20 mmHg | after 4, 8 weeks of treatment
Proportion of subjects achieving msitDBP < 90 mmHg and/or ΔmsitDBP ≥ 10 mmHg | after 4, 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Celltrion, Incheon, South Korea